CLINICAL TRIAL: NCT00783978
Title: Surfactant Disorders Associated With Chronic Lung Disease in Children.
Brief Title: Surfactant Disorders and Chronic Lung Disease
Acronym: APSE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM 07019
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Lung Disease
Keywords: Surfactant protein C; Interstitial; lung; Children

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, plasma, DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Children with chronic lung disease
  Interventions: Other: whole blood sample

INTERVENTIONS:
Other: whole blood sample — 2 ml of whole blood for children 5 ml of whole blood for parents that will be used only if 1 mutation is found in children

SUMMARY:
Interstitial lung diseases (ILD) in children represent a heterogeneous group of rare and not well defined disorders. Genetic abnormalities of surfactant proteins B (SFTPB) and more recently C (SFTPC) have been shown to be related to these pathologies. However, variability in the lung disease phenotype suggests the involvement of other surfactant-associated genes such as ABCA3 (ATP-binding cassette, sub-family A, member, 3). Thus, the aim of this project is: 1) to assess the prevalence of SFTPC mutation in children with chronic lung diseases, 2) to precise clinical and radiological features of children with SFTPC mutation, and 3) to identify environmental or genetic factors that may explain the extreme variability of this disease.

DETAILED DESCRIPTION:
The first stage of this project will be to constitute a clinical, radiological, biological database of children (1 moth-17 years) with severe respiratory distress and/or an unexplained chronic ILD. Mutations in SFTPC, SFTPB and ABCA3 will be further identified by sequencing and documented with using the parents blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Children from 1 month to 17 years old with radiological alveola-interstitial syndrome and:
* Oxygen weaning failure > 1 month in term newborn babies(>37th week of PCA)or> 40 weeks of PCA in preterm babies
* or
* Chronic respiratory disease define by chronic hypoxia and/or clinical signs of respiratory distress (cough, retractions, crackle)

Exclusion criteria:

* informed consent denied
* absence of social security

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: French pulmonary units participating to the study
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2009-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To assess the prevalence of SFTPC mutation in children with chronic lung diseases | At the inclusion visit

SECONDARY OUTCOMES:
To precise clinical and radiological features of children with SFTPC mutation | At the inclusion visit
To identify environmental or genetic factors that may explain the extreme variability of this disease | At the inclusion visit

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Epaud, MD, Principal Investigator — Hopital Trousseau, APHP
Locations (1):
- Hopital Trousseau, Paris, France

REFERENCES:
- [Derived] Epaud R, Delestrain C, Louha M, Simon S, Fanen P, Tazi A. Combined pulmonary fibrosis and emphysema syndrome associated with ABCA3 mutations. Eur Respir J. 2014 Feb;43(2):638-41. doi: 10.1183/09031936.00145213. Epub 2013 Oct 17. No abstract available. PMID 24136335
- [Derived] Delestrain C, Flamein F, Jonard L, Couderc R, Guillot L, Fanen P, Epaud R. [Lung diseases in children associated with inherited disorders of surfactant metabolism]. Rev Pneumol Clin. 2013 Aug;69(4):183-9. doi: 10.1016/j.pneumo.2013.05.002. Epub 2013 Jul 12. French. PMID 23856024
- [Derived] Flamein F, Riffault L, Muselet-Charlier C, Pernelle J, Feldmann D, Jonard L, Durand-Schneider AM, Coulomb A, Maurice M, Nogee LM, Inagaki N, Amselem S, Dubus JC, Rigourd V, Bremont F, Marguet C, Brouard J, de Blic J, Clement A, Epaud R, Guillot L. Molecular and cellular characteristics of ABCA3 mutations associated with diffuse parenchymal lung diseases in children. Hum Mol Genet. 2012 Feb 15;21(4):765-75. doi: 10.1093/hmg/ddr508. Epub 2011 Nov 7. PMID 22068586